CLINICAL TRIAL: NCT02022189
Title: Systematic Review of Clinical Biopsies of Dent Disease Patients
Brief Title: Review of Kidney Biopsies of Dent Disease Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, M.D., Mayo Clinic
Other Study IDs: 13-003738
Record Dates: First submitted 2013-12-06; First posted 2013-12-27 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Dent Disease
Keywords: Dent; Dents; Dent Disease; Renal Biopsy; Kidney Biopsy; Clinical Biopsy
MeSH Terms: conditions — Dent Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dent Disease patients: Patients with diagnosed Dent Disease
  Interventions: Procedure: Renal Biopsy

INTERVENTIONS:
Procedure: Renal Biopsy
  Other Names: All patients in the Dent Disease Registry with a previous renal biopsy.

SUMMARY:
This study is being done to obtain pathology reports from all patients in the Dent disease registry who have had a kidney biopsy. The investigator will collect the biopsy slides and reports in an attempt to determine if they have any common findings.

DETAILED DESCRIPTION:
If the patient agrees to be in the study, the patient will be asked to participate in the following:

* Sign a consent form indicating the patient's willingness to participate.
* Provide a signed medical release form allowing the investigator to request your official kidney biopsy reports, and also allowing the investigator to request the original slides for review. At the end of the study, all slides will be returned to the referring facility.
* The investigator will also review your medical record

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Dent Disease Registry with a previous renal biopsy.

Exclusion Criteria:

* None.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the Dent Registry with a previous renal biopsy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Biopsy changes | 2 years
  The primary outcome will be to determine the number of glomeruli, percent globally sclerotic glomeruli, percent focally sclerotic glomeruli, and the severity of interstitial fibrosis (none, mild, moderate, severe) and interstitial crystals (none, mild, moderate, severe)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Rare Kidney Stone Consortium — http://www.rarekidneystones.org